CLINICAL TRIAL: NCT04990817
Title: A Randomized, Controlled-feeding, Double-blind, Crossover Study to Examine the Metabolic Effects of Replacing Energy From Solid Fats and Added Sugars (SoFAS) With Avocado in Men and Women With Elevated Triglycerides
Brief Title: Effects of Replacing Energy From Solid Fats and Added Sugars (SoFAS) With Avocado
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Center for Metabolic and Cardiovascular Research (Other)
Collaborators: Hass Avocado Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MB-1914
Record Dates: First submitted 2021-07-26; First posted 2021-08-05 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Elevated Triglycerides; Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Average American Diet With SoFAS Replaced With Avocado (Experimental): Average American diet with foods that provide the equivalent of 1 medium to large avocado per day. It is anticipated that energy from avocado would replace 12-15% of daily energy, roughly half from solid fats and half from added sugars (SoFAS).
  Interventions: Other: Average American Diet With SoFAS Replaced With Avocado
- Average American Diet (Placebo Comparator): Average American diet based on macronutrient analyses from the most recent Nutrition and Health Examination Survey.
  Interventions: Other: Average American Diet

INTERVENTIONS:
Other: Average American Diet With SoFAS Replaced With Avocado — Replacing energy from solid fats and added sugars (SoFAS) with Avocado as part of an average American diet
  Arms: Average American Diet With SoFAS Replaced With Avocado
Other: Average American Diet — Average American diet based on macronutrient analyses from the most recent Nutrition and Health Examination Survey.
  Arms: Average American Diet

SUMMARY:
The objective of this study is to assess the effects of replacing energy from SoFAS with energy from avocado on non-high-density lipoprotein cholesterol (non-HDL-C) and other aspects of the cardiometabolic health profile including fasting lipoprotein lipid and particle concentrations, insulin sensitivity and blood pressure in men and women with elevated triglycerides (TG).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 21 to 74 y of age, inclusive.
2. Subject has a fasting fingerstick TG level of ≥135 mg/dL and <500 mg/dL at screening.
3. Subject has a BMI of 25.00 to 39.99 kg/m2, inclusive.
4. Subject has a vein access score of 7-10.
5. Subject is normally active and judged by the Investigator to be in general good health on the basis of medical history and screening measurements.
6. Subject is willing to comply with study food and background diet consumption during each treatment condition.
7. Subject is willing follow his/her regular physical activity pattern throughout the study period.
8. Subject is willing to refrain from consumption of all forms of recreational and/or medicinal marijuana (if legal) and alcoholic beverages for 24 h prior to each clinic visit requiring a blood draw.
9. Subject is willing to refrain from vigorous physical activity for 24 h prior to each clinic visit requiring a blood draw.
10. Subject is willing to abstain from caffeine use 1 h prior to and during each clinic visit
11. Subject is a non-smoker (at least 6 months), does not vape, and does not use other nicotine products and will abstain from use during the study period.
12. Subject who uses cannabidiol (CBD) and/or tetrahydrocannabinol (THC) has no plans to change habits during the study period.
13. Subject understands the study procedures and signs forms documenting informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator and is willing to complete study procedures.

Exclusion Criteria:

1. Subject has a laboratory test result of clinical significance based on the judgment of the Principal Investigator or qualified designee.
2. Subject has positive urine drug screen for illicit drugs.
3. Subject has fasting blood glucose ≥126 mg/dL at screening or known type 1 or type 2 diabetes mellitus.
4. Subject has atherosclerotic cardiovascular disease including any of the following: clinical signs of atherosclerosis including peripheral arterial disease, abdominal aortic aneurysm, carotid artery disease (symptomatic [e.g., myocardial infarction, angina, transient ischemic attack or stroke of carotid origin] or >50% stenosis on angiography or ultrasound) or other forms of clinical atherosclerotic disease (e.g., renal artery disease).
5. Subject has history or presence of a clinically significant gastrointestinal, endocrine, renal, hepatic, hematologic, immunologic, dermatologic, pulmonary, pancreatic, neurologic, psychiatric, inflammatory or biliary disorder that, in the opinion of the Investigator, could interfere with the interpretation of the study results.
6. Subject has a history of cancer in the prior 2 years, with the exception of non- melanoma skin cancer or carcinoma in situ of the cervix.
7. Subject has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg and/or diastolic blood pressure ≥100 mm Hg) at screening.
8. Subject has unstable use (defined as initiation or change in dose) of anti-hypertensive medication or thyroid hormone replacement within 4 weeks of screening.
9. Subject has used beta-adrenergic blockers and/or high-dose (>25 mg/d) thiazide diuretics within 4 weeks of screening.
10. Subject has unstable use (defined as initiation or change in dose, agent, or regimen) of statins within 4 weeks of screening.
11. Subject has used lipid-altering drugs other than statins including, but not limited to, bile acid sequestrants, cholesterol absorption inhibitors or fibrates within 4 weeks of screening.
12. Subject has used diabetes medications including alpha-glucosidase inhibitors, biguanides and biguanide combinations, thiazolidinediones, dipeptidyl peptidase-4 inhibitors, meglitinides and sulfonylureas and combination sulfonylureas within 4 weeks of screening.
13. Subject has used systemic corticosteroids within 4 weeks of screening.
14. Subject has used weight-loss drugs (including over-the-counter medications and/or supplements) or programs within 4 weeks prior to screening.
15. Subject has used lipid-altering foods, herbs or dietary supplements, including omega-3 fatty acid supplements with ≥900 mg/d EPA (eicosapentaenoic acid) or DHA (docosahexaenoic acid), niacin or its analogs at doses >200 mg/d, sterol/stanol products, dietary fiber supplements or red rice yeast supplements within 2 weeks of screening.
16. Subject has used dietary supplements that may affect carbohydrate metabolism, including chromium picolinate, ginseng, cinnamon (as a supplement) and starch blockers within 2 weeks of screening.
17. Subject has had a weight change of ±4.5 kg (10 lbs) in the previous 3 months.
18. Subject has an active infection and/or is on antibiotic therapy. Subject can be rescheduled for screening 7 days after completion of antibiotic therapy.
19. Subject has extreme dietary habits (e.g., vegan or very low carbohydrate diet).
20. Subject has a history of a diagnosed eating disorder (e.g., anorexia or bulimia nervosa).
21. Subject is a female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period.
22. Subject has a known allergy, sensitivity or intolerance to any foods.
23. Subject has been exposed to any non-registered drug product within 30 days of screening.
24. Subject has a current or recent history (past 12 months of screening) or strong potential for illicit drug or alcohol abuse. Alcohol abuse will be defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1.5 oz hard liquor).
25. Subject has a condition the Investigator believes would interfere with his or her ability to provide informed consent or comply with the study protocol, or which might confound the interpretation of the study results or put the person at undue risk.

Ages: 21 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
Non-HDL-C | Up to 21 days for each treatment period
  Percent change from baseline to the end of each treatment condition in non-HDL-C

SECONDARY OUTCOMES:
Total cholesterol (Total-C) | Up 21 days for each treatment period
  Change or percent change from baseline to the end of each treatment condition
High-density lipoprotein cholesterol (HDL-C) | Up to 21 days for each treatment period
  Change or percent change from baseline to the end of each treatment condition
Low-density lipoprotein cholesterol (HDL-C) | Up to 21 days for each treatment period
  Change or percent change from baseline to the end of each treatment condition
Triglyceride (TG) | Up to 21 days for each treatment period
  Change or percent change from baseline to the end of each treatment condition
Total-C/HDL-C Ration | Up to 21 days for each treatment period
  Change or percent change from baseline to the end of each treatment condition
Lipoprotein particle and subclass concentrations | Up to 21 days for each treatment period
  Change or percent change from baseline to the end of each treatment condition
Matsuda insulin sensitivity index | Up to 21 days for each treatment period
  Change or percent change from baseline to the end of each treatment condition
Disposition index from the liquid meal tolerance test [LMTT] (a measure of pancreatic beta-cell function) | Measured at baseline and end of each treatment period
  Change or percent change from baseline to the end of each treatment condition
Homeostasis model assessments of insulin sensitivity (HOMA2-%S), insulin resistance (HOMA-IR, linear model) and beta-cell function (HOMA2-%B) | Up to 21 days for each treatment period
  Change or percent change from baseline to the end of each treatment condition
Seated, resting systolic and diastolic blood pressures and heart rate | Up to 21 days for each treatment period
  Change or percent change from baseline to the end of each treatment condition

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Great Lakes Clinical Trials, Chicago, Illinois
  - I-CTSI Clinical Research Center, Indianapolis, Indiana

REFERENCES:
- [Derived] Gletsu-Miller N, Wilcox ML, Spence LA, Wright AJ, Guarneiri LL, Nadeem MM, Hutter MJ, Sprague KL, Brown AW, Friedman AN, Kirkpatrick CF, Maki KC. Effects of replacing solid fats and added sugars with avocado in adults with elevated cardiometabolic risk: a randomized, double-blind, controlled feeding, crossover trial. Am J Clin Nutr. 2025 Dec 13:101137. doi: 10.1016/j.ajcnut.2025.101137. Online ahead of print. PMID 41397527